CLINICAL TRIAL: NCT07319559
Title: Clinical Trial to Evaluate the Safety, Pharmacokinetic Characteristics of DW5124 and DW5124-R, and the Effect of Food on DW5124 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW5124-101
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R
- Sequence B (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R
- Sequence C (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R
- Sequence D (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R
- Sequence E (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R
- Sequence F (Experimental): cross-over
  Interventions: Drug: DW5124; Drug: DW5124-R

INTERVENTIONS:
Drug: DW5124 — DW5124 on fasted or fed condition
Drug: DW5124-R — DW5124-R on fasted or fed condition

SUMMARY:
This study aimed to evaluate the safety and pharmacokinetic characteristics of DW5124 and DW5124-R, and the effect of food on DW5124, in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers who are ≥19 years and >65 years old
* Body weight ≥50.0 kg and BMI between 18.0 and 30.0 kg/m2

Exclusion Criteria:

* Clinically significant Medical History
* In the case of women, pregnant(Urine-HCG positive) or lactating women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 72 hour
  Pharmacokinetics of DW5124-fed and DW5124-fasting, Pharmacokinetics of DW5124-fed and DW5124-R-fed
Area under the plasma concentration versus time curve (AUC) | up to 72 hour
  Pharmacokinetics of DW5124-fed and DW5124-fasting, Pharmacokinetics of DW5124-fed and DW5124-R-fed

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | up to 72 hour
  Pharmacokinetics of DW5124-fed, DW5124-fasting, DW5124-R-fed
Terminal half life (t1/2) | up to 72 hour
  Pharmacokinetics of DW5124-fed, DW5124-fasting, DW5124-R-fed
Apparent clearance (CL/F) | up to 72 hour
  Pharmacokinetics of DW5124-fed, DW5124-fasting, DW5124-R-fed
Apparent volume of distribution (Vd/F) | up to 72 hour
  Pharmacokinetics of DW5124-fed, DW5124-fasting, DW5124-R-fed

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea